CLINICAL TRIAL: NCT00391768
Title: A Pharmacokinetic/Pharmacodynamic and Safety Evaluation of Oseltamivir (Tamiflu®) for the Treatment of Children Less Than 24 Months of Age With Confirmed Influenza Infection (CASG 114)
Brief Title: Oseltamivir Treatment for Children Less Than 24 Months of Age With Influenza
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0059; N01AI30025C; Roche WP-20749; CASG 114; N01AI30025 (NIH)
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Results first posted 2011-06-20 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2010-02

CONDITIONS: Influenza
Keywords: influenza, oseltamivir, Tamiflu®, antiviral, children, infants
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (1):
- oseltamivir (Tamiflu®) (Experimental)
  Interventions: Drug: oseltamivir (Tamiflu®)

INTERVENTIONS:
Drug: oseltamivir (Tamiflu®) — Oseltamivir is supplied as a white powder blend for constitution to a suspension. It is supplied in 100 ml amber glass bottles with 30 grams of powder for oral suspension, a plastic adapter, a plastic oral dispenser and a plastic measuring cup. Initially subjects in Cohort I received oseltamivir 30 mg orally twice daily for 5 days. The DSMB recommended on 05-Aug-2009 that weight based dosing of oseltamivir for subjects subsequently enrolled in Cohort I. Based on pharmacokinetic data available as of that date, the initial weight-based dose to be evaluated for Cohort I is 3.5 mg/kg twice a day. Cohort II and Cohort III will receive oseltamivir at 3.0 mg/kg/dose orally twice daily for 5 days. Cohorts IV and V will receive 3.0 mg/kg/dose orally twice daily for 5 days, this dose may be adjusted.

SUMMARY:
The purpose of this study is to learn how to treat influenza in children less than 2 years of age. Tamiflu®, the drug being studied, is approved for treatment of children 1 year of age and older with influenza. Researchers want to learn more about the activity of Tamiflu® in the body to determine a dose of that is safe, well-tolerated, and effective in young children with influenza. Children less than 24 months of age with confirmed influenza will receive Tamiflu® 2 times a day for 5 days. Older participants will be enrolled first and younger children will be enrolled after the safety data is reviewed for older participants. Study procedures include blood samples, swabs from inside the nose, and body and nervous system evaluations. Participants may be involved in study related procedures for up to 37 days.

DETAILED DESCRIPTION:
Oseltamivir is approved for prophylaxis and treatment of children 1 year of age and older with influenza. Influenza treatments for children under the age of 1 year are needed because mortality from influenza is high among this age group, even when there are no underlying medical conditions. Oseltamivir is frequently used off-label in children less than 1 year of age, with no data supporting the doses being used. Given the risk of severe or fatal influenza infection in infants, the lack of repeat dose pharmacokinetic (PK) data in children less than 2, the need for treatments in this population of children, and the fact that oseltamivir is being used off-label in this population, the current study will systematically study the PK and safety of oseltamivir in children less than 2 years of age with confirmed influenza to determine the appropriate dose to be used in these age groups. This data will be critical to pediatricians caring for these potentially gravely ill infants. This study is a prospective, age-stratified PK/pharmacodynamic (PD) and safety evaluation of oseltamivir therapy in children less than 24 months of age with confirmed influenza infection. Participants will be stratified by age into the following enrollment scheme at study initiation: 12-23 months (Cohort I), 9-11 months (Cohort II), 6-8 months (Cohort III), 3-5 months (Cohort IV) and 0-2 months (Cohort V). At study onset, Cohort II and III will be enrolled simultaneously. Cohorts IV and V will be enrolled sequentially by decreasing age groups predicated upon the PK and safety data from the preceding cohort. In the event of a public health emergency, the Data Safety Monitoring Board (DSMB) or Food and Drug Administration (FDA) may authorize the following modifications to the proposed enrollment plan: the opening of younger age cohorts without the full dataset from the next higher age cohort, the re-opening of previously closed cohorts to obtain additional data and/or the over-enrollment of any of the 5 cohorts. The oldest cohort (Cohort I) may be enrolled at any time during the study. The primary study objective is to define the PK of oseltamivir and oseltamivir carboxylate in children with confirmed influenza less than 2 years of age. The oseltamivir dose initially evaluated in Cohort I was the approved dose of 30 mg twice a day (bid). However, the oseltamivir carboxylate area under the curve (AUC)12 values for 5 of the 9 subjects enrolled in Cohort I as of August 5, 2009, were below the lower range utilized for the other cohorts in the study, as was the GM AUC12 for Cohort I as a group [(2589 nanograms per hour per milliliter (ngxh/mL)]. As a consequence, the DSMB recommended on August 5, 2009, that the protocol be amended to utilize weight-based dosing of oseltamivir in subjects subsequently enrolled in Cohort I, and to employ the targeted AUC approach used for Cohorts II-V for this cohort as well. Based upon the PK data available as of that date, the initial weight-based dose to be evaluated for Cohort I is 3.5 mg/kg bid. A dose of oseltamivir 3 mg/kg/dose orally bid for 5 days (10 doses) will be administered to the first 9 subjects in each of Cohorts II-III. Additional subjects may be enrolled if the target AUC12 range is not achieved. The proposed dose for subjects enrolled in Cohorts IV and V will be 3 mg/kg/dose orally bid for 5 days (10 doses), although this dose may be adjusted prior to opening Cohort IV or V based on the dose required to achieve the target oseltamivir carboxylate AUC12 range in the previous cohort.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s).
* Age:

Cohort I: 12 - 23 mo. Cohort II: 9 - 11 mo. Cohort III: 6 - 8 mo. Cohort IV: 3 - 5 mo. Cohort V: 0 - 2 mo.

* Confirmed laboratory diagnosis of influenza by viral culture or rapid influenza diagnostic test within 96 hours prior to study enrollment.
* Duration of influenza symptoms less than or equal to 96 hours.

Exclusion Criteria:

* Concomitant vomiting illness that would preclude ability to take drug.
* Immunocompromised subject (e.g., malignancy, congenital agammaglobulinemia, HIV).
* Documented renal impairment (e.g., polycystic renal disease, nephrectomy, renal transplantation, renal agenesis, dialysis requirement, renal failure, nephrotic syndrome at any time prior to enrollment, current receipt of diuretic therapy).
* Documented hepatic impairment (e.g., congenital hepatitis, biliary atresia, cholelithiasis).
* Gastrointestinal abnormality which might hinder absorption of an oral medication.
* Current receipt of inotropic drugs (e.g., epinephrine, norepinephrine, dopamine, dobutamine).
* History of seizures.
* Documented congenital malformations of the central nervous system defined at birth (e.g., hydranencephaly, prosencephaly, spina bifida).

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arkansas Children's Hospital - Infectious Diseases, Little Rock, Arkansas
  - Miller Children's Hospital Long Beach - Bickerstaff Family Center, Long Beach, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado - Infectious Disease, Aurora, Colorado
  - Children's National Medical Center - Sheikh Zayed Campus - Infectious Disease, Washington D.C., District of Columbia
  - University of Florida - Shands Children's Hospital, Gainesville, Florida
  - University of South Florida - Tampa General Hospital - Pediatrics, Tampa, Florida
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Emory University School of Medicine - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Louisiana State University Health Shreveport - Pediatrics, Shreveport, Louisiana
  - University of Mississippi - Children's Infectious Diseases, Jackson, Mississippi
  - Washington University School of Medicine in St. Louis - Center for Clinical Studies, St Louis, Missouri
  - University of Nebraska Medical Center - Children's Hospital and Medical Center - Infectious Diseases, Omaha, Nebraska
  - Cohen Children's Medical Center - Pediatric Infectious Diseases, Manhasset, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - MetroHealth Medical Center - Pediatric Infectious Disease, Cleveland, Ohio
  - Children's Hospital of Philadelphia - The Center for Pediatric Clinical Effectiveness, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC - General Academic Pediatric, Pittsburgh, Pennsylvania
  - Rhode Island Hospital - Pediatrics, Providence, Rhode Island
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Infectious Disease Services, Fort Worth, Texas
  - University of Utah - Pediatric Pharmacology Program, Salt Lake City, Utah
  - Seattle Children's Hospital - Infectious Diseases, Seattle, Washington
- Canada (3):
  - University of Alberta Hospital - Pediatrics, Edmonton, Alberta
  - The Hospital for Sick Children - Infectious Diseases, Toronto, Ontario
  - Centre Hospitalier de l'Universite Laval/ CHUQ, Québec, Quebec

REFERENCES:
- [Result] Kimberlin DW, Acosta EP, Prichard MN, Sanchez PJ, Ampofo K, Lang D, Ashouri N, Vanchiere JA, Abzug MJ, Abughali N, Caserta MT, Englund JA, Sood SK, Spigarelli MG, Bradley JS, Lew J, Michaels MG, Wan W, Cloud G, Jester P, Lakeman FD, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Oseltamivir pharmacokinetics, dosing, and resistance among children aged <2 years with influenza. J Infect Dis. 2013 Mar 1;207(5):709-20. doi: 10.1093/infdis/jis765. Epub 2012 Dec 10. PMID 23230059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the emergency department, hospital, physician's office or clinical care unit. Children of both sexes and all races were included. The recruitment period was January 2007 through May 2010.
Groups:
- Cohort IA: 12 - 23 months of age, 30 mg
- Cohort IB: 12 - 23 months of age, 3.5 mg/kg body weight
- Cohort IIA: 9 - 11 months of age, 3 mg/kg body weight
- Cohort IIB: 9 to 11 months of age, 3.5 mg/kg body weight
- Cohort III: 6 to 8 months of age, 3 mg/kg body weight
- Cohort IV: 3 to 5 months of age, 3 mg/kg body weight
- Cohort V: 0 to 2 months of age, 3 mg/kg body weight
Period: Overall Study
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Started | 12 | 3 | 7 | 8 | 24 | 10 | 23
Completed | 12 | 3 | 6 | 7 | 22 | 7 | 19
Not Completed | 0 | 0 | 1 | 1 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V | Total
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23 | 87
Age, Customized [Number; unit: Participants] | 12 | 3 | 7 | 8 | 24 | 10 | 23 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 6 | 13 | 2 | 8 | 36
  Male | 9 | 2 | 4 | 2 | 11 | 8 | 15 | 51
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 7 | 8 | 24 | 10 | 23 | 87

OUTCOME MEASURES:

1. Primary Outcome: Oseltamivir Carboxylate AUC12 (Area Under the Curve).
Description: The oseltamivir carboxylate AUC12 was derived from a series of five blood draws over 10 to 12 hours.
Time Frame: Day 3 of drug administration
Population: Subjects that received 3 days study drug administration and had successful PK draws on study day 3.
Measure: Number; unit: participants
Groups:
- Cohort IA: Subjects aged 12 to 23 months of age confirmed to have influenza. These subjects received 30mg of Oseltamivir twice a day times 5 days.
- Cohort IB: Subjects 12 to 23 months of age confirmed to have influenza and received 3.5 mg/kg of Oseltamivir by mouth twice a day times 5 days.
- Cohort IIA: Subjects 9 to 11 months of age confirmed to have influenza and received 3 mg/kg body weight of Oseltamivir by mouth twice a day times 5 days.
- Cohort IIB: Subjects 9 to 11 months of age confirmed to have influenza and received 3.5 mg/kg body weight of Oseltamivir by mouth twice a day times 5 days.
- Cohort III: Subjects 6 to 8 months of age confirmed to have influenza and received 3 mg/kg body weight of Oseltamivir by mouth twice a day times 5 days.
- Cohort IV: Subjects 3 to 5 months of age confirmed to have influenza and received 3 mg/kg body weight of Oseltamivir by mouth twice a day times 5 days.
- Cohort V: Subjects 0 to 2 months of age confirmed to have influenza and received 3 mg/kg body weight of Oseltamivir by mouth twice a day times 5 days.
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 10 | 3 | 6 | 7 | 22 | 10 | 19
participants
  AUC12 <2660 | 6 | 1 | 3 | 0 | 2 | 0 | 3
  AUC12 > or = 2660 and <7700 | 4 | 2 | 3 | 7 | 19 | 10 | 13
  AUC12 > or =7700 | 0 | 0 | 0 | 0 | 1 | 0 | 3

2. Secondary Outcome: Overall Reported Adverse Events (AEs) Thought to be Associated With Study Therapy.
Description: Any event considered associated with drug that occurred post first dose of drug administration that was not present at baseline was considered an AE. Expected flu symptoms were not reported as AEs but were collected separately.
Time Frame: Duration of study, from receipt of the first dose of study drug and continuing through study visit Day 30 plus or minus 3 days.
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Groups:
- Cohort IA: Subjects aged 12 - 23 months of age confirmed to have influenza. These subjects received 30 mg of Oseltamivir twice a day times 5 days.
- Cohort IB: Subjects aged 12 - 23 months of age confirmed to have influenza. These subjects received 3.5 mg/kg body weight of Oseltamivir twice a day times 5 days.
- Cohort IIA: Subjects aged 9 - 11 months of age confirmed to have influenza. These subjects received 3 mg/kg body weight of Oseltamivir twice a day times 5 days.
- Cohort IIB: Subjects aged 9 - 11 months of age confirmed to have influenza. These subjects received 3.5 mg/kg body weight of Oseltamivir twice a day times 5 days.
- Cohort III: Subjects aged 6 - 8 months of age confirmed to have influenza. These subjects received 3 mg/kg body weight of Oseltamivir twice a day times 5 days.
- Cohort IV: Subjects aged 3 - 5 months of age confirmed to have influenza. These subjects received 3 mg/kg body weight of Oseltamivir twice a day times 5 days
- Cohort V: Subjects aged 0 - 2 months of age confirmed to have influenza. These subjects received 3 mg/kg body weight of Oseltamivir twice a day times 5 days
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23
participants
  Event - Vomiting | 3 | 0 | 0 | 0 | 2 | 0 | 0
  Event - Dermatitis Diaper | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Event - Rash | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Number and Characteristics of Adverse Events (AEs) Described as Neurological Events.
Description: Any neurological event that occurred post first dose of drug administration that was not present at baseline was considered an AE. Expected flu symptoms were not reported as AEs but were collected separately.
Time Frame: as for outcome 2
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23
participants
  Event - Lethargy | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Event - Tremor | 0 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Incidence of Treatment Emergent AEs and Drug Related AEs by Cohort and Toxicity Grade
Description: Any event considered to be related to the study drug that occurred post first dose of drug administration that was not present at baseline was considered an AE. Expected flu symptoms were not reported as AEs but were collected separately. The Division of AIDS Toxicity Tables (DIAIDS) were used to grade the events.
Time Frame: as for outcome 2
Population: Intention to treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23
Participants
  Grade I - Mild | 3 | 0 | 0 | 0 | 3 | 0 | 1
  Grade II - Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade III - Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade IV - Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade V - Death | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Incidence of Treatment Emergent AEs and Drug Related AEs by Cohort Leading to Discontinuation of Study Medication
Description: Study drug was administered for 5 days; any event that occurred prior to the last dose of study medication that was considered related to an AE and that caused the subject to stop taking study drug.
Time Frame: Duration of study, from receipt of the first dose of study drug and continuing through study visit Day 5 plus or minus 1 day
Measure: Number; unit: events
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23
events | 0 | 0 | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Incidence of All Serious Adverse Events by Cohort and System Organ Class (SOC)
Description: Serious Adverse Event (SAE) were classified by MedDRA System Organ Class (SOC). An SAE was reported if it met the following criteria and occurred after the first dose of study medication through the end of the study: death throughout study participation; life threatening; requires inpatient hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance; results in congenital anomaly or birth defect; results in a persistent or significant disability; and an event considered serious by the PI.
Time Frame: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 12 | 3 | 7 | 8 | 24 | 10 | 23
Participants
  Total | 2 | 0 | 1 | 2 | 2 | 1 | 0
  General Disorders & Administration Site Conditions | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Immune System Disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Infections and Infestations | 2 | 0 | 0 | 1 | 1 | 0 | 0
  Investigations | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory, thoracic & mediastinal disorders | 0 | 0 | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Correlation of Clearance of Viral RNA by Culture With Pharmacokinetic Parameters by Cohort
Description: The Spearman coefficient and the p-values were computed between the clearance of Viral RNA and Oseltamivir Carboxylate Area under the curve from 0 to 12 hours (AUC0-12)
Time Frame: Day to negative viral load for subjects positive at baseline
Population: Subjects included in this analysis are those who had positive culture at baseline (day 0) and had a negative culture on one of the following study visit days: Day 3, Day 5 or Day 10. Culture was obtained from a a nasal swab. Subjects also would have had evaluable PK samples on study day 3.
Measure: Number; unit: Spearman coefficient
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 8 | 2 | 4 | 5 | 12 | 8 | 18
Spearman coefficient | 0.67 | NA — too few subjects | 0.40 | 0.62 | 0.09 | 0.30 | 0.01
Statistical Analysis 1: Comparison: Cohort IA; Test type: Superiority or Other; p = 0.07, Spearman Correlation
Statistical Analysis 2: Comparison: Cohort IIA; Test type: Superiority or Other; p = 0.60, Spearman Correlation
Statistical Analysis 3: Comparison: Cohort IIB; Test type: Superiority or Other; p = 0.27, Spearman Correlation
Statistical Analysis 4: Comparison: Cohort III; Test type: Superiority or Other; p = 0.77, Spearman Correlation
Statistical Analysis 5: Comparison: Cohort IV; Test type: Superiority or Other; p = 0.47, Spearman Correlation
Statistical Analysis 6: Comparison: Cohort V; Test type: Superiority or Other; p = 0.96, Spearman Correlation

8. Secondary Outcome: Correlation of Clearance of Viral RNA by Polymerase Chain Reaction (PCR) to Pharmacokinetic Parameters by Cohort.
Description: The Spearman coefficient and the p-values were computed between the clearance of viral RNA and oseltamivir carboxylate Area Under the Curve from 0 to 12 hours (AUC 0-12)
Time Frame: From date of enrollment until the date of first documented absence of viral load by culture, assessed up to 10 days after enrollment.
Population: Subjects included in this analysis are those who had viral loads at baseline (day 0) and had a non-detectable viral load on one of the following study visit days: day 3, day 5, or day 10. Virus was obtained from a nasal swab. Subjects also would have had evaluable PK samples on study day 3.
Measure: Number; unit: correlation measure
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Number analyzed (Participants) | 10 | 2 | 4 | 5 | 16 | 8 | 18
correlation measure
  AUC0-12 (hr*ng/mL) unit: Spearman Coefficient | 0.57 | NA — too few subjects available | 0.21 | 0.90 | 0.28 | 0.04 | 0.07
  AUC0-12 (hr*ng/mL) unit: P value | 0.08 | NA — too few subjects available | 0.79 | 0.04 | 0.30 | 0.93 | 0.77

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were collected from Day 1 to Day 30 of protocol
Arm/Group | Cohort IA | Cohort IB | Cohort IIA | Cohort IIB | Cohort III | Cohort IV | Cohort V
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/3 | 1/7 | 2/8 | 2/24 | 1/10 | 0/23
Other Adverse Events (participants affected / at risk) | 8/12 | 1/3 | 3/7 | 6/8 | 18/24 | 3/10 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort IA (N=12) | Cohort IB (N=3) | Cohort IIA (N=7) | Cohort IIB (N=8) | Cohort III (N=24) | Cohort IV (N=10) | Cohort V (N=23)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pnuemonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort IA (N=12) | Cohort IB (N=3) | Cohort IIA (N=7) | Cohort IIB (N=8) | Cohort III (N=24) | Cohort IV (N=10) | Cohort V (N=23)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida nappy rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No